CLINICAL TRIAL: NCT05345301
Title: Electroencephalographic Correlates of Glove-stretch Therapy Post-stroke
Brief Title: Safety and Feasibility of eGlove
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, James Patton, Director, Robotics Laboratory, Arms and Hands Lab, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU00216276
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Stroke
Keywords: Upper Extremity; Body Computer Interface
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Measuring neural activity (Experimental): While completing hand opening/closing, individuals will have the following measured (1) Neural activity (specifically sensorimotor rhythms) using a EEG cap; (2) muscle activity (specifically finger flexors and extensors) using EMG sensors.
  Interventions: Diagnostic Test: Event related desynchronization measurement

INTERVENTIONS:
Diagnostic Test: Event related desynchronization measurement — Individuals will spend one hour and receive cues to open or close their hand while wearing a EEG cap and EMG sensors on their forearm.

SUMMARY:
The purpose of this study is to measure how cortical signals improve in stroke participants after passive hand stretching therapy from a robotic glove.

DETAILED DESCRIPTION:
After experiencing a stroke event, many individuals are left with life-long motor impairments in their upper extremity. However, motor recovery for stroke survivors is not fully understood. One of the challenges to understand the mechanisms behind recovery is the capability of the brain to reorganize and re-activate areas affected by the stroke. Brain computer interface (BCI) has shown promise in previous studies to improve motor capabilities of individuals with damaged nervous systems by reactivating damaged motor pathways.

In order to understand how BCI can be incorporated into upper extremity rehabilitation, investigators must first lay the groundwork of measuring neural activity and its relation to muscle activity in individuals who have experienced a stroke. While instructing participants to open and close their hand, investigators will measure (1) neural activity, called sensorimotor rhythms (SMRs), using a electrophysiological (EEG) cap, and (2) muscle activity using wireless electromyography (EMGs). What the investigators are specifically looking for is an event in the neural activity in between movement initiation and termination called event related desynchronization (ERD). The investigators of this study hypothesize that there is greater activation of ERDs in stroke's subjects SMR activity after completing finger extension and flexion.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke (6 months post stroke)
* Hemiparesis
* Some degree of hand and finger movement capability
* a moderate impairment (Fugl-Meyer score between 15-50)

Exclusion Criteria:

* Individuals under the age of 18
* Bilateral paresis
* Hand pain and/or extreme articular contractures on the finger joints (Modified Ashworth Scale of 4)
* Botox injection to the affected upper extremity within the previous 4 months
* Aphasia, cognitive impairment, or affective dysfunction that would influence the ability to perform the experiment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Rate of activation of Event Related Desynchronization | 1 hour
  Sensorimotor neural activity

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

REFERENCES:
- [Result] Ang KK, Guan C, Chua KS, Phua KS, Wang C, Chin ZY, Zhou L, Tang KY, Joseph GJ, Kuah C. A clinical study of motor imagery BCI performance in stroke by including calibration data from passive movement. Annu Int Conf IEEE Eng Med Biol Soc. 2013;2013:6603-6. doi: 10.1109/EMBC.2013.6611069. PMID 24111256
- [Result] Buch E, Weber C, Cohen LG, Braun C, Dimyan MA, Ard T, Mellinger J, Caria A, Soekadar S, Fourkas A, Birbaumer N. Think to move: a neuromagnetic brain-computer interface (BCI) system for chronic stroke. Stroke. 2008 Mar;39(3):910-7. doi: 10.1161/STROKEAHA.107.505313. Epub 2008 Feb 7. PMID 18258825
- [Result] Dobkin B, Barbeau H, Deforge D, Ditunno J, Elashoff R, Apple D, Basso M, Behrman A, Harkema S, Saulino M, Scott M; Spinal Cord Injury Locomotor Trial Group. The evolution of walking-related outcomes over the first 12 weeks of rehabilitation for incomplete traumatic spinal cord injury: the multicenter randomized Spinal Cord Injury Locomotor Trial. Neurorehabil Neural Repair. 2007 Jan-Feb;21(1):25-35. doi: 10.1177/1545968306295556. PMID 17172551
- [Result] Peles O, Werner-Reiss U, Bergman H, Israel Z, Vaadia E. Phase-Specific Microstimulation Differentially Modulates Beta Oscillations and Affects Behavior. Cell Rep. 2020 Feb 25;30(8):2555-2566.e3. doi: 10.1016/j.celrep.2020.02.005. PMID 32101735
- [Result] Triandafilou KM, Kamper DG. Carryover effects of cyclical stretching of the digits on hand function in stroke survivors. Arch Phys Med Rehabil. 2014 Aug;95(8):1571-6. doi: 10.1016/j.apmr.2014.04.008. Epub 2014 May 2. PMID 24794423
- [Result] Thielbar KO, Triandafilou KM, Fischer HC, O'Toole JM, Corrigan ML, Ochoa JM, Stoykov ME, Kamper DG. Benefits of Using a Voice and EMG-Driven Actuated Glove to Support Occupational Therapy for Stroke Survivors. IEEE Trans Neural Syst Rehabil Eng. 2017 Mar;25(3):297-305. doi: 10.1109/TNSRE.2016.2569070. Epub 2016 May 17. PMID 27214905
- [Result] McFarland DJ, Sarnacki WA, Wolpaw JR. Effects of training pre-movement sensorimotor rhythms on behavioral performance. J Neural Eng. 2015 Dec;12(6):066021. doi: 10.1088/1741-2560/12/6/066021. Epub 2015 Nov 3. PMID 26529119
- [Result] Ramos-Murguialday A, Broetz D, Rea M, Laer L, Yilmaz O, Brasil FL, Liberati G, Curado MR, Garcia-Cossio E, Vyziotis A, Cho W, Agostini M, Soares E, Soekadar S, Caria A, Cohen LG, Birbaumer N. Brain-machine interface in chronic stroke rehabilitation: a controlled study. Ann Neurol. 2013 Jul;74(1):100-8. doi: 10.1002/ana.23879. Epub 2013 Aug 7. PMID 23494615
- [Result] Seo NJ, Rymer WZ, Kamper DG. Delays in grip initiation and termination in persons with stroke: effects of arm support and active muscle stretch exercise. J Neurophysiol. 2009 Jun;101(6):3108-15. doi: 10.1152/jn.91108.2008. Epub 2009 Apr 8. PMID 19357330
- [Result] Yuan H, He B. Brain-computer interfaces using sensorimotor rhythms: current state and future perspectives. IEEE Trans Biomed Eng. 2014 May;61(5):1425-35. doi: 10.1109/TBME.2014.2312397. PMID 24759276
- [Result] Prasad G, Herman P, Coyle D, McDonough S, Crosbie J. Applying a brain-computer interface to support motor imagery practice in people with stroke for upper limb recovery: a feasibility study. J Neuroeng Rehabil. 2010 Dec 14;7:60. doi: 10.1186/1743-0003-7-60. PMID 21156054
- [Result] Morone NE, Greco CM, Moore CG, Rollman BL, Lane B, Morrow LA, Glynn NW, Weiner DK. A Mind-Body Program for Older Adults With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA Intern Med. 2016 Mar;176(3):329-37. doi: 10.1001/jamainternmed.2015.8033. PMID 26903081